CLINICAL TRIAL: NCT02330042
Title: Functional Optical Coherence Tomography-Derived Biomarkers for Diabetic Retinopathy
Brief Title: OCT Biomarkers for Diabetic Retinopathy
Status: Active, not recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Thomas Hwang, MD, Professor of Ophthalmology, Retina & Vitreous Diseases Division, Oregon Health and Science University
Other Study IDs: IRB#00010949
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes; OCT; Angiography; Diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Patients with:
  * Type 1 or Type 2 diabetes mellitus
  * severe non-proliferative diabetic retinopathy (NPDR) or proliferative diabetic retinopathy (PDR).
- Group B: Patients with:
  * Type 1 or Type 2 diabetes mellitus
  * with or without mild to moderate NPDR
- Group C (controls): Patients without diabetes or evidence of any form of eye disease

SUMMARY:
Diabetic retinopathy (DR) is caused by changes in the blood vessels of the retina associated with long-term Type 1 or Type 2 diabetes mellitus. DR is a leading cause of blindness in the United States. Standard optical coherence tomography (OCT) cannot directly detect vascular changes, which may occur early affecting the passage of blood through the tiny capillaries (reduced capillary flow) or cause the greatest damage through formation of abnormal blood vessel growth (neovascularization). Currently, fluorescein angiography (FA) is the gold standard for detecting these changes, but FA requires an injection of a dye into the vein of the arm of the patient. This dye can cause undesirable side effects. Recently, OCT has been used to make functional measurements (such as total retinal blood flow among others) and to perform angiography. Thus, functional OCT may provide a useful, alternate way to evaluate diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria for participants with diabetes:

* Male or female participants 18-79 years old
* With Type 1 diabetes for over 5 years or Type 2 diabetes of any duration

Exclusion Criteria for participants with diabetes:

* Vision worse than 20/200
* Inability to maintain fixation for OCT imaging
* Significant kidney disease, kidney failure or kidney transplant
* Unstable medical status, including blood pressure greater than 180/110 or unstable heart disease
* Pregnant or nursing an infant
* Presence of an eye disease (other than diabetic retinopathy) that can affect retinal blood flow, retinal permeability or retinal anatomy
* Significant cataract, corneal scar, vitreous bleed or other media opacity
* History of major eye surgery within 4 months prior to enrollment in this study

Inclusion Criteria for participants without diabetes (controls):

* Male or female participants 18-79 years old

Exclusion Criteria for participants without diabetes (controls):

* Vision worse than 20/200
* Inability to maintain fixation for OCT imaging
* Significant kidney disease, kidney failure or kidney transplant
* Unstable medical status, including blood pressure greater than 180/110 or unstable heart disease
* Pregnant or nursing an infant
* Presence of any eye disease that can affect retinal blood flow, retinal permeability or retinal anatomy
* Significant cataract, corneal scar, vitreous bleed or other media opacity
* History of major eye surgery within 4 months prior to enrollment in this study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with Type 1 diabetes of greater than 5 years duration OR Type 2 diabetes of any duration. Healthy controls are also being enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with decreased total retinal blood flow by OCT angiography | 1 year
  Total retinal blood flow will be measured in uL/min.
Number of participants with capillary dropout and/or new abnormal retinal blood vessel growth by OCT angiography | 1 year
  Neovascular membrane area will be measured in mm2.
Number of participants with measureable macular edema by OCT imaging | 1 year
  Retinal thickening area will be measured in mm2.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hwang, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States